CLINICAL TRIAL: NCT06962969
Title: Real-world Database Study to Observe Safety and Effectiveness of Ibrance
Brief Title: A Study to Understand the Patients Confirmed to Have Advanced or Metastatic Breast Cancer and Receiving Palbociclib Treatment Using a Real-world Database
Status: Not yet recruiting | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A5481186
Record Dates: First submitted 2025-04-30; First posted 2025-05-08 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Advanced or Metastatic Breast Cancer
Keywords: breast cancer; Palbociclib
MeSH Terms: conditions — Breast Neoplasms | interventions — palbociclib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Ibrance (palbociclib): Patients who received at least one initial prescription of Ibrance following a diagnosis of advanced/metastatic breast cancer
  Interventions: Drug: Ibrance

INTERVENTIONS:
Drug: Ibrance — Patients who received at least one initial prescription of Ibrance following a diagnosis of advanced/metastatic breast cancer
  Other Names: Palbociclib

SUMMARY:
The purpose of this real-world study is to look at breast cancer patients receiving Palbociclib using a large real-world database collected under real-world practice. This study also looks at the safety of Ibrance, including any side effects. Side effects are undesired effects of a medicine or other type of treatment.

This study will include the data of the following participants:

* Adult women (more than18 years of age) with at least one visit with a breast cancer
* Patients with locally advanced breast cancer or metastatic breast cancer with a staging classification of stage III, stage IV. Advanced cancer is a term that is often used to describe cancer that is unlikely to be cured. Metastatic cancer is the cancer which is spread from the place where it started to other places in the body.
* Patients with a laboratory test positive for hormone receptor and negative for HER2 before or up to 60 days after advanced/metastatic breast cancer diagnosis date.
* Patients who received at least one initial prescription of Ibrance following a diagnosis of advanced/metastatic breast cancer.

This study will look at the safety of palbociclib treatment by looking at the number and severity of the side effects.

ELIGIBILITY:
Inclusion Criteria

Patients must meet all of the following inclusion criteria to be eligible for inclusion in the study:

* Adult women (≥ 18 years of age) with at least one visit with a breast cancer ICD10 diagnosis code (C50.x)
* Patients with locally advanced breast cancer or metastatic breast cancer with a staging classification of stage III, stage IV (distant metastases).
* Patients with a laboratory test positive for hormone receptor (HR) and negative for human epithelial growth factor receptor 2 (HER2) before or up to 60 days after advanced/metastatic breast cancer diagnosis date.

  1. HR-positive is defined as any positive test for estrogen receptor or progesterone receptor.
  2. HER2-negative is defined as any HER2-negative test and the absence of a positive test (immunohistochemistry positive (3+), fluorescence in situ hybridization positive/amplified).
* Patients who received at least one initial prescription of Ibrance following a diagnosis of advanced/metastatic breast cancer

Exclusion Criteria

Patients meeting any of the following criteria will not be included in the study:

* Breast cancer with HR-negative and HER2-positive on laboratory testing.
* More than a 90-day gap between breast cancer diagnosis date and next visit.
* Patients who treated as off-label

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study participants will be patients diagnosed with HR(+)/HER2(-) advanced/metastatic breast cancer between August 29, 2015 and September 30, 2023 who meet the general prescribing criteria for Palbociclib in South Korea according to the national product manual, and who meet the following inclusion and exclusion criteria, as determined by data from one year prior to the Ibrance approval date
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-06-30 (Estimated); Primary Completion 2025-11-28 (Estimated); Study Completion 2025-11-28 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events that occur during treatment | From index date to last dose plus 28 days. Index is defined as the date of first prescription of Ibrance on participants diagnosed between 29 Aug 2015 through 30 Sep 2023
Number of participants with associated risk factors | From index date to last dose plus 28 days. Index is defined as the date of first prescription of Ibrance on participants diagnosed between 29 Aug 2015 through 30 Sep 2023

SECONDARY OUTCOMES:
Overall Survival (OS) | From baseline to the date of death or censoring date, whichever occurs first on participants diagnosed between 29 Aug 2015 through 30 Sep 2023
Real-World Tumor Response (rwTR) | From baseline to the date of death or censoring date, whichever occurs first on participants diagnosed between 29 Aug 2015 through 30 Sep 2023

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.